CLINICAL TRIAL: NCT05239793
Title: Translational Studies on Electronic Cigarette-derived Oxidants and Their Long-term Cardiopulmonary Effects
Brief Title: Electronic Cigarette-derived Oxidants and Cardiopulmonary Effects
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Rebecca Bascom, Professor, Department of Medicine, Penn State Health Milton S Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00015514; 1R01HL152436 (NIH)
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NJOY e-cigarette (Other): NJOY e-cigarette containing 5% nicotine strength pods
  Interventions: Drug: NJOY e-cigarette

INTERVENTIONS:
Drug: NJOY e-cigarette — NJOY e-cigarette with Virginia Tobacco flavored 5% nicotine pods

SUMMARY:
This is a pilot study on the impact of switching from cigarettes to Electronic Cigarettes (EC) on disease-related clinical symptoms and biomarkers of harm in smokers with preexisting Chronic Obstructive Pulmonary Disease (COPD). The researchers hypothesize that the smokers who switch to EC completely or significantly will experience reduced COPD symptoms, risks of exacerbations, and decreased levels of oxidative stress and inflammation.

DETAILED DESCRIPTION:
Smokers with COPD have a higher pack-year history and nicotine dependence compared to regular smokers as exemplified by the relatively large proportion of patients diagnosed with COPD that continue to smoke (95%).

This is a translational project which addresses the changing profile of tobacco product use in the United States (US) and the need for data regarding toxicity pathways for new nicotine products such as EC. In particular it focuses on critical scientific and clinically relevant gaps relating to oxidants in EC and their potential long-term cardiopulmonary effects. The study will obtain new information regarding the potential cardiopulmonary toxicity resulting from exposure to EC-derived oxidants that may lead to long-term disease development.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate COPD
* Smokes a popular brand of cigarette
* Willing to use an e-cigarette to reduce cigarette smoking down to 75% of their daily baseline cigarette use
* Ability to read, write and understand English
* Ability to provide informed consent and attend study visits

Exclusion Criteria:

* History of active, chronic drug abuse or alcohol abuse problems
* Actively changing smoking behavior
* Unwilling or unable to provide blood samples
* Pregnant, planning to become pregnant, or nursing
* Use of tobacco products other than cigarettes in the past 30 days
* Recent history (< 6 months) of myocardial infarction (MI)
* Any unstable or life threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or drug therapy within the past year. Antiarrhythmic drugs include amiodarone, flecainide, IV ibutilide, IV lidocaine, procainamide, propafenone, quinidine, tocainide
* Hospitalization for heart failure (NY Heart Association III or IV) within the past year
* Uncontrolled hypertension
* Known allergy to vegetable glycerin and propylene glycol
* History of seizures or medications to prevent seizures

Ages: 21 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cigarettes per day | 3 months
  Self reported cigarettes per day
Number of exacerbations | 3 months
  Number of COPD exacerbations

SECONDARY OUTCOMES:
Lung function tests (spirometry) | 3 months
  FEV1
COPD Assessment Test (CAT) scores | 3 months
  8-item scale with range of scores from 0-40. Higher scores denote a more severe impact of COPD on a patient's life.
6-min walk distance (6MWD) | 3 months
  This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes.
Tobacco exposure | 3 months
  Measure by cotinine (ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Bascom, MD, Principal Investigator — Penn State Health Hershey Medical Center; Raghu Sinha, PhD, Principal Investigator — Penn State Health Hershey Medical Center
Locations (1):
- Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We propose to make de-identified data, codebooks, documentation, and research protocols available to interested researchers after completion of the study.
Supporting Information: Study Protocol
Time Frame: Data will be available within 3 years of the culmination of data collection activities.
Access Criteria: Any investigator interested in collaboration or in using the data collected in this study for their own work will be invited to submit a 1-page abstract of their proposed research, including purpose, analytical plan, and dissemination plans. The study leadership team will review these proposals and decide on each based on the individual merits. Review criteria and prioritization of projects include: potential of the proposed work to advance public health, qualifications of the applicant, the potential for publication, the potential for future funding, and enhancing the scientific, geographic, and demographic diversity of the research portfolio.